CLINICAL TRIAL: NCT03668769
Title: Project Quitting Schedule
Brief Title: Quitting Schedule Mobile Smartphone Application in Helping Participants to Quit Smoking
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: 0 participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0516; NCI-2018-01820 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0516 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Cigarette Smoker; Current Every Day Smoker; Current Smoker; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic; Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (smoking reduction, Quitting Schedule mobile app) (Experimental): AIM I: Participants follow an individually tailored gradual reduction of smoking schedule for 5 weeks while MDACC eHealth adapts WebCASSI into a smartphone app: Quitting Schedule.
  AIM II: Participants pre-test the Quitting Schedule mobile smartphone app for 5 weeks.
  Interventions: Other: Internet Mobile Technology; Other: Interview; Other: Questionnaire Administration; Behavioral: Smoking Cessation Intervention

INTERVENTIONS:
Other: Internet Mobile Technology — Use Quitting Schedule mobile smartphone app
  Other Names: www-mobile
Other: Interview — Ancillary studies
Other: Questionnaire Administration — Ancillary studies
Behavioral: Smoking Cessation Intervention — Participate in individual smoking cessation program
  Other Names: Smoking and Tobacco Use Cessation Interventions

SUMMARY:
This trial studies how well a mobile smartphone application called Quitting Schedule works in helping participants to quit smoking. Quitting Schedule is based on WebCASSI, a computer-based initiative that offered state of-the-art smoking cessation treatment and counseling to MD Anderson Cancer Center (MDACC) patients and served as a portal for non-patients to find information regarding smoking cessation advice and treatments. Quitting Schedule may help participants to quit smoking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To adapt the internal algorithms of the scheduled reduced smoking approach in Computer Assisted Stop Smoking Intervention for the World Wide Web (WebCASSI) into a smartphone application (app): Quitting Schedule.

II. Once the smartphone app is developed, a pretesting phase with smoker seeking care at MDACC Tobacco Treatment Program or another community service such as Equality Texas, Lesbian, Gay, Bisexual, Transgender, and Queer (LGBTQ) Advisory Board of the City of Houston, Montrose Center, Avenue 360 and Lesbian Health Initiative will follow.

III. To culturally and linguistically adapt Quitting Schedule app into Spanish language.

IV. To implement a feasibility trial in IDC (Colombia), INCan (Mexico), and INEN (Peru).

OUTLINE:

AIM I: Participants follow an individually tailored gradual reduction of smoking schedule for 5 weeks while MDACC eHealth adapts WebCASSI into a smartphone app: Quitting Schedule.

AIM II: Participants pre-test the Quitting Schedule mobile smartphone app for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Current smokers (those who smoke at least 5 cigarettes a day; confirmed with carbon monoxide (CO) levels equal or above 7 parts per million ) newly enrolled in the Tobacco Treatment Program at MDACC (Aim 2 )
* Male or female (Aim 2)
* Adult cancer patients - 18 years or older (Aim 2)
* Current smokers seeking care at the Tobacco Treatment Program at MD Anderson and at Houston area community services who have smoked at least 100 cigarettes in lifetime
* Willing to download and use the app Quitting Schedule (Aim 2)
* Willing to set a quit smoking date within 5 weeks of the enrollment (Aim 2)
* Ownership of an iPhone or Android smartphone (Aim 2)

Exclusion Criteria:

* Unwillingness to participate in the study (Aim 2)
* Enrolled in another cessation program (Aim 2)
* Current use of NRT or other smoking cessation medications,e.g. Varenicline or Bupropion outside of the MD Anderson Institution (Aim 2)
* Expired CO levels below 7ppm (Aim 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Adaptation of the programmatic infrastructure of WebCASSI (Computer Assisted Stop Smoking Intervention for the World Wide Web) into a more-portable table and smartphone application (app) that will be available both in English and Spanish | Up to 5 weeks
Pre-testing of the app | Up to 5 weeks
  A focus group will be used in order to provide feedback on the features of the app in relation to usability for smoking cessation and future app development.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cinciripini, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org